CLINICAL TRIAL: NCT03920033
Title: Comparison of Salvage Hypofractionated Accelerated Versus Standard Radiotherapy for Biochemical Recurrence After Radical Prostatectomy (SHARE Trial): a Prospective, Randomized Controlled, Open-label, Multi Center, Superiority Study
Brief Title: Salvage Hypofractionated Accelerated Versus Standard Radiotherapy for Biochemical Failure After Prostatectomy
Acronym: SHARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young Seok Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2019-0154-0001
Record Dates: First submitted 2019-03-25; First posted 2019-04-18 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer; Biochemical Recurrence; Radiation; Hypofractionation; Dose Escalation; Survival; Radiation Toxicity; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated (Experimental): 65 Gy/ 26 fractions (fraction size 2.5 Gy)
  Interventions: Radiation: Salvage radiation therapy
- Standard (Active Comparator): 66 Gy/ 33 fractions (fraction size 2 Gy)
  Interventions: Radiation: Salvage radiation therapy

INTERVENTIONS:
Radiation: Salvage radiation therapy — Salvage radiation therapy for biochemical recurrence

SUMMARY:
Patients with a biochemical recurrence after radical prostatectomy for moderate- or high- risk prostate cancer are randomly assigned to hypofractionated, accelerated high dose radiation therapy group (65 Gy, 26 fractions) and a control group of standard treatment group (66 Gy, 33 fractions). The criteria for stratification at randomization include 1) risk groups, 2) androgen deprivation therapy, and 3) PSA before salvage radiation therapy, which affect biochemical recurrence.

It is expected that hypofractionated, accelerated high dose radiation therapy will have a superiority in terms of biochemical control to conventional radiation therapy, and the present study would like to confirm this. In addition, we aimed to evaluate and compare the toxicity and quality of life index of two radiation therapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed intermediate- or high-risk prostate cancer
* Biochemical recurrence after radical prostatectomy (Definition: Serial elevation of PSA over 0.2 ng/mL and <=1.0 ng/mL)
* ECOG performance status 0-1
* Appropriate values of blood tests within 6 months after enrollment Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 Platelets ≥ 50,000 cells/mm3 Hemoglobin ≥ 8.0 g/dl
* Appropriate values of kidney function within 6 months after enrollment Creatinine < 2.0 ng/dL
* Appropriate values of liver function within 6 months after enrollment total bilirubin < 1.5 X maximum normal value alanine aminotransferase or aspartate aminotransferase < 2.5 X maximum normal value

Exclusion Criteria:

* Clinically gross recurrent tumor
* Presence of distant metastasis
* Presence of pelvic LN metastasis
* History of pelvic irradiation
* History of cryotherapy or brachytherapy for prostate cancer
* Double primary cancer other than skin/thyroid cancer
* Combined serious morbidity

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence-free survival | 5 years
  PSA >0.2 ng/mLfollowed by a repeat measurement >0.2 ng/mL

SECONDARY OUTCOMES:
Acute toxicities | Adverse effects occured during radiation therapy, and within 3 months after radiation therapy
  Evaulation using CTCAE 4.0 Evaluation using CTCAE 4.0 CTCAE 4.0
Chronic toxicities | Adverse effects occured after 3 months since end of radiation therapy
  Evaulation using CTCAE 4.0
Quality of life 1 | the date of enrollment, up to 1 week after radiation therapy, 6 months, every year until 5 years
  Expanded prostate cancer index composite (EPIC) Questionnaire Korean version EPIC consists of 50 questions in total divided into four domains: bowel (14 questions), urinary (12 questions), sexual (13 questions), and hormonal aspects (13 questions).
  Scores of each domain will be separately reported. Response options for each EPIC item form a Likert scale, and multi-item scale scores will be summed and transformed linearly to a 0-to-100 scale.
  The higher the score, the higher the quality of life.
Quality of life 2 | the date of enrollment, up to 1 week after radiation therapy, 6 months, every year until 5 years
  European Organization for Research and Treatment Core Quality of Life Questionnaire (EORTC QLQ-C30) Korean version EORTC QLQ-C30 consists of 30 questions, and total score will be reported. Response options for each EPIC question form a Likert scale, and multi-item scale scores will be summed and transformed linearly to a 0-to-100 scale.
  The higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Young Seok Kim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Park G, Kim YJ, Ahn H, Park W, Lee JS, Kim YS. Salvage hypofractionated accelerated versus standard radiotherapy for the treatment of biochemical recurrence after radical prostatectomy (SHARE): the protocol of a prospective, randomized, open-label, superiority, multi-institutional trial. Trials. 2021 Oct 21;22(1):728. doi: 10.1186/s13063-021-05708-5. PMID 34674739